CLINICAL TRIAL: NCT05691101
Title: Comparison of Quality of Recovery in Patients Using Continuous Brachial Plexus Block With or Without Intravenous Patient-Controlled Analgesia After Arthroscopic Rotator Cuff Repair: A Prospective Randomized Study
Brief Title: Comparison of Using CIBPB With or Without IV-PCA After Arthroscopic Rotator Cuff Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Ji In Park, Principal Investigator, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: B-2210/789-001
Record Dates: First submitted 2023-01-10; First posted 2023-01-19 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Analgesia, Patient-Controlled; Brachial Plexus Block; Arthroscopic Rotator Cuff Repair
Keywords: Postoperative pain; IV PCA; Continuous interscalene brachial plexus block
MeSH Terms: conditions — Agnosia; Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous interscalene brachial plexus block(CISB) with IV PCA group (Experimental): Patients in this group received continuous interscalene brachial plexus block(CISB) and intravenous PCA
  Interventions: Other: CISB with IV PCA group
- Continuous interscalene brachial plexus block (CISB) group (Active Comparator): Patients in this group received continuous interscalene brachial plexus block (CISB)
  Interventions: Other: CISB group

INTERVENTIONS:
Other: CISB with IV PCA group — Ultrasonography guided interscalene brachial plexus block was done with a 5 cm block needle and catheter was inserted. (Stimuplex®A, B Braun Medical, Bethlehem, PA). 10 mL 0.375 % ropivacaine was injected through the catheter.
  0.2 % ropivacaine 4 ml/hour was injected through the continuous brachial plexus block catheter. IV-PCA with fentanyl (basal flow 0 ml with patient selected bolus 14 mcg, lockout 10 minutes) was started.
  Arms: Continuous interscalene brachial plexus block(CISB) with IV PCA group
Other: CISB group — Ultrasonography guided interscalene brachial plexus block was done with a 5 cm block needle and catheter was inserted. (Stimuplex®A, B Braun Medical, Bethlehem, PA). 10 mL 0.375 % ropivacaine was injected through the catheter.
  0.2 % ropivacaine (4 ml/hour with patient selected bolus 5 ml, lockout 60 minutes) was injected through the continuous brachial plexus block catheter.
  Arms: Continuous interscalene brachial plexus block (CISB) group

SUMMARY:
The goal of this study is to compare the continuous brachial plexus block with or without intravenous patient controlled analgesia(PCA) in patients undergoing arthroscopic rotator cuff repair, in terms of quality of recovery, postoperative pain score, and adverse event.

DETAILED DESCRIPTION:
The Bellomic® M silicone balloon infuser, dual continuous petite type (cebika, Uiwang-si, Gyeonggi-do, Republic of Korea) has 2-channel infusion elastomeric pump with two balloon chambers.

This structure allows the simultaneous use of continuous nerve block and intravenous PCA. In addition, intravenous PCA can be continued even when continuous nerve block is discontinued due to discomfort such as numbness, tingling sense or motor block.

This is expected to contribute to the patient satisfaction and quality of recovery.

ELIGIBILITY:
Inclusion Criteria:

* Having arthroscopic rotator cuff repair
* American Society of Anesthesiologists physical status I-III

Exclusion Criteria:

* Contraindication to interscalene brachial plexus block
* Contraindication to fentanyl

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-01-31 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Korean version of the Quality of Recovery-15 questionnaire (QoR-15K) score (0-150, 0: poor recovery, 150: good recovery) | Postoperative 24 hour
  Patient recovery measured by QoR-15K score

SECONDARY OUTCOMES:
Pain score | Postoperative 6, 24, 48 hour
  Numerical Rating Scale (NRS-11(0-10): 0:no Pain and 10:Severe/Worst Pain)
Cumulative consumption of PCA and rescue analgesics | Postoperative 24, 48 hour
  Cumulative consumption of systemic analgesics
Occurrence of adverse effects | Postoperative 24, 48 hour
  Nausea, vomiting, numbness, tingling sense, motor and sensory blockade

CONTACTS AND LOCATIONS:
Overall Officials: JI IN PARK, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul national univercity Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No